CLINICAL TRIAL: NCT04122976
Title: Darolutamide Observational Study in Non-metastatic Castration-resistant Prostate Cancer Patients
Brief Title: A Study in Which Non-metastatic Castration-resistant Prostate Cancer (nmCRPC) Patients for Whom a Decision to Treat With Darolutamide Has Been Made Before Enrollment Are Observed and Certain Outcomes Are Described
Acronym: DAROL
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20590
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with nmCRPC: Men with nmCRPC for whom a decision to treat with darolutamide has been made before enrollment, and who have signed informed consent, will be eligible for the study.
  Interventions: Drug: Darolutamide(Nubeqa, BAY1841788)

INTERVENTIONS:
Drug: Darolutamide(Nubeqa, BAY1841788) — The decision on the dose and duration of treatment is solely at the discretion of the treating physician, based on the recommendations written in the local product information.

SUMMARY:
The purpose of this study is to find out in the real-world setting, if darolutamide is safe and effective for patients diagnosed with prostate cancer that has not spread to other parts of the body. When a patient is enrolled to the study, his/her physician would have already made the decision to treat patient with darolutamide per local standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of 18 years
* Histologically or cytologically confirmed adenocarcinoma CRPC defined by disease progression despite ADT and may present as a confirmed rise in serum PSA levels (as defined by PCWG3: Rising PSA values at a minimum of 1-week intervals, and a baseline PSA value ≥ 1.0 ng/mL). For patients with a prior ARi treatment (Enzalutamide or Apalutamide), there is no baseline PSA value required
* No evidence of metastasis based on conventional imaging. An imaging assessment needs to be obtained prior to the 1st dose of darolutamide. For patients with a prior ARi treatment (Enzalutamide or Apalutamide) for nmCRPC, M0 status with no evidence of disease progression should be confirmed within 3 months of ARi discontinuation
* Decision to initiate treatment with darolutamide was made as per investigator's routine treatment practice prior to enrollment in the study
* Signed informed consent
* Life expectancy of ≥3 months
* For a patient with a prior ARi treatment (Enzalutamide or Apalutamide) for nmCRPC for less than one year, all toxic effects from prior use of any ARi treatment have to be resolved at the time of enrollment and prior to the 1st dose of darolutamide

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Contraindications according to the local marketing authorization
* Previous treatment with darolutamide (more than 3 days prior to enrollment)
* Patient with a prior ARi treatment (Enzalutamide or Apalutamide) for nmCRPC for more than one year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with a diagnosis of nmCRPC will be enrolled after the decision for treatment with darolutamide has been made by the investigator.
Sampling Method: Non-Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse events (TEAEs) | Up to 30 days after last dose of darolutamide within the patient's observation period
  Including severity, seriousness and outcome.
Reasonable causal relationship between darolutamide and an adverse event (AE) | Up to 30 days after last dose of darolutamide within the patient's observation period
Action taken related to darolutamide treatment | Up to 30 days after last dose of darolutamide within the patient's observation period
  Dose modifications and time periods

SECONDARY OUTCOMES:
Subject's demographics | Up to 7 years
Subject's characteristics | Up to 7 years
Co-morbidities | Up to 7 years
Disease course and progression (including performance status) | Up to 7 years
Concomitant medication/treatment (including opioids) | Up to 7 years
Dosage and dose modification of darolutamide | Up to 7 years
Reasons for ending treatment and/or observation/follow-up | Up to 7 years
Metastasis-Free Survival (MFS) | Up to 7 years
Time to Symptomatic Skeletal Event (TSSE) | Up to 7 years
Time to Prostate-Specific Antigen (PSA) progression | Up to 7 years
Survival rate | Up to 7 years
Duration of darolutamide therapy | Up to 7 years
Imaging exams used to define tumor status | Up to 7 years
Imaging exams (as chosen by treating physician) used to diagnose nmCRPC (including date and clinical finding) | Up to 7 years
Prior and post - darolutamide treatments for prostate cancer | Up to 7 years

CONTACTS AND LOCATIONS:
Locations (41):
- United States (25):
  - Urology Centers of Alabama, Homewood, Alabama
  - Arizona Institute of Urology, Tucson, Arizona
  - Genesis Comprehensive Prostate Cancer Center, San Diego, California
  - The Urology Center of Colorado, Denver, Colorado
  - Manatee Medical Research Institute, Bradenton, Florida
  - Advanced Urology Institute, Daytona Beach, Florida
  - Research by Design, LLC, Chicago, Illinois
  - First Urology, PSC, Jeffersonville, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - Southcoast Centers for Cancer Care, Fairhaven, Massachusetts
  - New Jersey Urology, Englewood, New Jersey
  - Beacon Cancer Care, Beacon, New York
  - Integrated Medical Professionals, PLLC, North New Hyde Park, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Associated Medical Professional Urology, Syracuse, New York
  - Dukes Cancer Intitute Center for Prostate and Urologic Cancers, Durham, North Carolina
  - Associated Urologists of NC, Raleigh, North Carolina
  - Oregon Urology Institutue, Springfield, Oregon
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology San Antonio, San Antonio, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - Urology of Virginia, Virginia Beach, Virginia
  - University of Washington, Seattle, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Many Locations, Multiple Locations, Argentina
- Many Locations, Multiple Locations, Austria
- Many Locations, Multiple Locations, Belgium
- Many Locations, Multiple Locations, Brazil
- Many Locations, Multiple Locations, Canada
- Many Locations, Multiple Locations, China
- Many Locations, Multiple Locations, Colombia
- Many Locations, Multiple Locations, Denmark
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Greece
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Japan
- Many Locations, Multiple Locations, Russia
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.